CLINICAL TRIAL: NCT01099904
Title: The Effect of Renal Function on the Pharmacokinetics of RO4995855 (Parent of ProDrug RO5024048) Following Multiple Oral Dose Administration of RO5024048
Brief Title: A Study on the Effect of Renal Function on the Pharmacakokinetics of RO5024048 (Parent of Prodrug RO5024048) Following Multiple Oral Dose Administration of RO5024048
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: PP21536
Record Dates: First submitted 2010-04-06; First posted 2010-04-08 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

ARMS (3):
- 1 (Experimental): Normal Renal Function
  Interventions: Drug: RO5024048
- 2 (Experimental): Mild Renal Impairment
  Interventions: Drug: RO5024048
- 3 (Experimental): Moderate Renal Impairment
  Interventions: Drug: RO5024048

INTERVENTIONS:
Drug: RO5024048 — multiple oral doses for 5 days

SUMMARY:
This open-label, parallel group study will evaluate the effect of renal function on the pharmacokinetics of RO4995855 following multiple oral dose administration of RO5024048 and assess the effect of renal impairment on safety and tolerability of RO5024048. Adult males or females with either normal renal function or mild or moderate renal impairment will receive RO5024048 orally for 5 days. Target sample size is <50.

ELIGIBILITY:
Inclusion Criteria:

* male or female adults, 18-75 years of age
* normal, or mildly or moderately impaired renal function (creatinine clearance >/= 30 mL/min)
* BMI 18-40 kg/m2
* stable renal function
* agree to abstain from alcohol consumption during study drug adminsitration and limit consumption up to the end of the study
* agree to abstain from coffein consumption throughout study

Exclusion Criteria:

* positive urine or blood test for drugs of abuse not under a physician's prescription
* positive for HIV or HCV, or HBV with clinical symptoms or history of hepatitis
* uncontrolled hypertension
* renal transplant, dialysis patient, nephritic syndrome
* clinically significant cardiovascular, central nervous system, gastrointestinal or liver disease or disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Phrmacokinetics of RO49958855 (parent molecule) and metabolites following multiple doses of RO5024048: AUC, Cmax, Tmax T1/2, Ae, Cl | sampling days 1 and 3-11

SECONDARY OUTCOMES:
Effect of renal impairment on safety and tolerability: Adverse events, vital signs, ECG, laboratory parameters | Throughout study, ECG and laboratory assessments days 3, 5, 6 and 17

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- United States (2):
  - Orlando, Florida
  - Knoxville, Tennessee
- Christchurch, New Zealand